CLINICAL TRIAL: NCT03709680
Title: PHASE 1/2 STUDY TO EVALUATE PALBOCICLIB (IBRANCE®) IN COMBINATION WITH IRINOTECAN AND TEMOZOLOMIDE OR IN COMBINATION WITH TOPOTECAN AND CYCLOPHOSPHAMIDE IN PEDIATRIC PATIENTS WITH RECURRENT OR REFRACTORY SOLID TUMORS
Brief Title: Study Of Palbociclib Combined With Chemotherapy In Pediatric Patients With Recurrent/Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5481092; 2024-511975-14-00 (Registry Identifier: CTIS (EU))
Expanded Access: Available
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Ewing Sarcoma; Solid Tumors; Rhabdoid Tumor; Rhabdomyosarcoma; Neuroblastoma; Medulloblastoma; Diffuse Intrinsic Pontine Glioma
Keywords: Ewing Sarcoma; EWS; Neuroblastoma; Recurrent Neuroblastoma; Solid Tumor; Recurrent Solid Tumors; Refractory Solid Tumors; Bone Cancer; Bone Tumor; Bone Sarcoma; Soft Tissue Cancer; Soft Tissue Sarcoma; Recurrent Ewing Sarcoma; Refractory Ewing Sarcoma; Relapsed Ewing Sarcoma; Pediatric Cancer; Childhood Cancer; Ewing Sarcoma Treatment; Palbociclib; CDK4/6 Inhibitor; Irinotecan; Temozolomide; Topotecan; Cyclophosphamide
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdoid Tumor; Rhabdomyosarcoma; Neuroblastoma; Medulloblastoma; Diffuse Intrinsic Pontine Glioma; Bone Neoplasms; Sarcoma; Neoplasms | interventions — palbociclib; Temozolomide; Irinotecan; Topotecan; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Phase 1 portion: The palbociclib plus irinotecan and temozolomide combination part of the study will comprise of a dose escalation cohort (following a rolling 6 design), a dose expansion cohort.
  The palbociclib plus topotecan and cyclophosphamide will comprise of a dose determination cohort(following a modified rolling 6 design), a dose expansion cohort, and Neuroblastoma tumor -specific cohort.
  Phase 2 open-label, randomized portion of the study will randomize patients in a 2:1 ratio to receive either palbociclib in combination with irinotecan and temozolomide (Arm A) or irinotecan and temozolomide chemotherapy alone (Arm B). Randomization will be stratified using block randomization by type and time of current disease recurrence (primary refractory or 1st recurrence < 2 years versus 1st recurrence ≥ 2 years or 2nd or greater recurrence).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Phase 2 Arm A (Experimental): Palbociclib in combination with irinotecan and temozolomide.
  Interventions: Drug: Palbociclib; Drug: Temozolomide; Drug: Irinotecan
- Phase 1 (Experimental): Palbociclib in combination with temozolomide and irinotecan and/or with topotecan and cyclophosphamide.
  Interventions: Drug: Palbociclib; Drug: Temozolomide; Drug: Irinotecan; Drug: Topotecan; Drug: Cyclophosphamide
- Phase 2 Arm B (Active Comparator): Irinotecan and temozolomide alone.
  Interventions: Drug: Temozolomide; Drug: Irinotecan
- Phase 1 Tumor specific cohort - Neuroblastoma (Experimental): Palbociclib in combination with topotecan and cyclophosphamide.
  Interventions: Drug: Palbociclib; Drug: Topotecan; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Palbociclib — Phase 1: Administered (oral) at 55 mg/m2, 75 mg/m2, or 40 mg/m2, or 95 mg/m2 or 115 mg/m2 on days 1-14 of a 21-day cycle Phase 1 Tumor specific cohort-Neuroblastoma and Phase 2 : Administered (oral) at 75 mg/m2 on days 1-14 of a 21-day cycle
  Other Names: Ibrance
  Arms: Phase 1; Phase 1 Tumor specific cohort - Neuroblastoma; Phase 2 Arm A
Drug: Temozolomide — Phase 1 and Phase 2: Administered at 100 mg/m2 (oral or intravenous), on days 1-5 of a 21-day cycle
  Other Names: Temodar
  Arms: Phase 1; Phase 2 Arm A; Phase 2 Arm B
Drug: Irinotecan — Phase 1 and Phase 2: Administered at 50 mg/m2 (intravenous), on days 1-5 of a 21-day cycle
  Other Names: Campto
  Arms: Phase 1; Phase 2 Arm A; Phase 2 Arm B
Drug: Topotecan — Phase 1 only : Administered at 0.75 mg/m2 (intravenous), on days 1-5 of a 21-day cycle
  Other Names: Hycamtin
  Arms: Phase 1; Phase 1 Tumor specific cohort - Neuroblastoma
Drug: Cyclophosphamide — Phase 1 only: Administered at 250 mg/m2 (intravenous), on days 1-5 of a 21-day cycle
  Other Names: Cytoxan
  Arms: Phase 1; Phase 1 Tumor specific cohort - Neuroblastoma

SUMMARY:
A study to learn about safety and find out maximum tolerable dose of palbociclib given in combination with chemotherapy (temozolomide with irinotecan or topotecan with cyclophosphamide) in children, adolescents and young adults with recurrent or refractory solid tumors (phase 1). Neuroblastoma tumor specific cohort to further evaluate antitumor activity of palbociclib in combination with topotecan and cyclophosphamide in children, adolescents, and young adults with recurrent or refractory neuroblastoma. Phase 2 to learn about the efficacy of palbociclib in combination with irinotecan and temozolomide when compared with irinotecan and temozolomide alone in the treatment of children, adolescents, and young adults with recurrent or refractory Ewing sarcoma (EWS).

ELIGIBILITY:
Inclusion:

1. Histologically confirmed relapsed or refractory solid tumor as follows:

   * For dose escalation and dose determination parts: Histologically confirmed relapsed or refractory solid tumor (including CNS tumors but not lymphomas). Patients with Diffuse Intrinsic Pontine Glioma do not require histological only radiographic confirmed relapse to enroll.
   * For dose expansion and tumor specific cohorts: Histologically confirmed relapsed or refractory solid tumor including but not limited to EWS, rhabdoid tumor, rhabdomyosarcoma, neuroblastoma, and medulloblastoma. Patients with Diffuse Intrinsic Pontine Glioma do not require histological only radiographic confirmed relapse to enroll. EWS is not eligible for TOPO and CTX tumor-specific cohorts.
   * For randomized Phase 2 part: Histologically confirmed Ewing sarcoma at diagnosis or at relapse, with presence of EWSR1-ETS or FUS-ETS rearrangement. Histopathology confirmation of both EWSR1-ETS or FUS-ETS rearrangement partners is required OR availability of formalin fixed paraffin embedded (FFPE) tumor tissue sample for central testing. Patient must have relapsed or have refractory disease and at least evaluable disease in at least one site other than bone marrow that can be followed by imaging.
2. Age ≥2 and <21 years at the time of study entry.
3. Lansky performance status ≥50% for patients ≤16 years of age, or Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2 for patients >16 years of age.
4. Adequate bone marrow function.

   * Absolute neutrophil count ≥1000/mm3;
   * Platelet count ≥75,000/mm3 (transfusion independent, no platelet transfusion in past 7 days prior study entry);
   * Hemoglobin ≥8.5 g/dL (transfusion allowed).
5. Adequate renal function: Serum creatinine level based on age/gender must within protocol specified limits.
6. Adequate liver function, including:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)

     ≤2.5 × upper limit of normal (ULN) or ≤5 × ULN for age, if attributable to disease involvement of the liver;
   * Total bilirubin ≤1.5 × ULN for age, unless the patient has documented Gilbert's syndrome.Patients with documented Gilbert's syndrome are eligible if direct bilirubin is within normal ranges (≤ULN).
7. Patients enrolled to Phase 1 portion of the study and tumor specific cohorts must have measurable disease as defined by RECIST version 1.1 or modified RANO criteria for CNS disease or at least evaluable disease by INRC for neuroblastoma.

   The eligible patients with neuroblastoma must have at least one of the following at the time of study entry:
   * Measurable tumor by CT or MRI that is avid on MIBG scan or demonstrates increased FDG uptake on PET scan;
   * Avid lesion on MIBG scan with positive uptake at a minimum of one site;
   * For disease that is not avid by MIBG-scan, at least one lesion that demonstrates increased FDG uptake on PET scan AND viable neuroblastoma confirmed by current or prior biopsy;
   * bone marrow involvement with more than 5% neuroblastoma cells in at least one sample from bilateral bone marrow biopsies;
   * In non MIBG-avid refractory soft tissue disease that does not demonstrate increased FDG uptake; lesion biopsy is required to document the presence of viable neuroblastoma, unless patient has a new soft tissue lesion (radiographic evidence of disease progression).

   Patients with EWS enrolled to Phase 2 portion of the study are eligible with evaluable disease (eg, bone only disease with no soft tissue component).
8. Recovered to CTCAE Grade ≤1, or to baseline, from any non-hematological acute toxicities of prior surgery, chemotherapy, immunotherapy, radiotherapy, differentiation therapy or biologic therapy, with the exception of alopecia.
9. Serum/urine pregnancy test (for all girls ≥8 years of age) negative at screening and at the baseline visit.

Exclusion:

1. Phase 1 and tumor specific cohorts: For palbociclib with IRN and TMZ combination, prior treatment with a CDK4/6 inhibitor or progression while on treatment with an IRN-containing regimen that includes TMZ. Patients who have received the combination of IRN and TMZ and did not progress while on these medications are eligible. For patients enrolling in the palbociclib with TOPO and CTX combination, prior treatment with a CDK4/6 inhibitor or progression while on treatment with a TOPO-containing regimen that includes CTX. Patients who have received the combination of TOPO and CTX and did not progress while on these medications are eligible. Phase 2 portion: prior treatment with a CDK4/6 inhibitor or progression while on treatment with an IRN-containing or TMZ-containing regimen. Patients who have received IRN and/or TMZ and did not progress while on these medications are eligible.
2. Prior intolerability to IRN and/or TMZ plus/minus palbociclib with IRN and TMZ combination and prior intolerability to TOPO and/or CTX for TOPO and CTX combination. For patients enrolled in the UK, any contraindication for IRN and/or TMZ treatment, as per the local SmPC.
3. Use of strong cytochrome P450 (CYP) 3A inhibitors or inducers within 12 days of study entry. Patients who are receiving strong uridine diphosphate-glucuronosyl transferase 1A1 (UGT1A1) inhibitors within 12 days of Cycle 1 Day 1 (C1D1) are not eligible for the palbociclib with IRN and TMZ combination. Patients who are receiving strong UGT1A1 inhibitors within 12 days of C1D1 are eligible for the palbociclib with TOPO and CTX combination (See Section 5.7.1 for list of products.)
4. Systemic anti cancer therapy within 2 weeks prior to study entry and 6 weeks for nitrosoureas.
5. Prior irradiation to >50% of the bone marrow (see Appendix 9).
6. Participation in other studies involving investigational drug(s) within 2 weeks or 5 half lives, whichever is longer, prior to study entry.
7. Major surgery within 4 weeks prior to study entry. Surgical biopsies or central line placement are not considered major surgeries.
8. For IRN and TMZ with/without palbociclib combinations: known or suspected hypersensitivity to palbociclib, dacarbazine, IRN and/or TMZ. For combination of palbociclib with TOPO and CTX: known or suspected hypersensitivity to palbociclib, TOPO and/or CTX.
9. Patients with known symptomatic brain tumors or brain metastases and require steroids, unless they have been on a stable or on a decreasing steroid dose for >14 days.
10. Patients with previously diagnosed brain metastases are eligible if they have completed their prior treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry for these metastases for at least 14 days post radiation and 4 weeks post-surgery and are neurologically stable.
11. Hereditary bone marrow failure disorder.
12. QTc >470 msec.
13. History of clinically significant or uncontrolled cardiac disease, including:

    * History of or active congestive heart failure; if patient had congestive heart failure resolve and >1 year from resolution, patient will be considered eligible;
    * Clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation or Torsades de Pointes);
    * Diagnosed or suspected congenital or acquired prolonged QT syndrome;
    * Need for medications known to prolong the QT interval;
    * Uncorrected hypomagnesemia or hypokalemia because of potential effects on the QT interval;
    * Left ventricular ejection fraction <50% or shortening fraction <28%.
14. Recent or ongoing clinically significant gastrointestinal disorder that may interfere with absorption of orally administered drugs (eg, gastrectomy).
15. Evidence of serious active or uncontrolled bacterial, fungal or viral infection or known history of hepatitis B virus, hepatitis C virus, or human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness. Screening for viral hepatitis and HIV is under discretion of investigator unless required by local regulation.
16. Severe acute or chronic medical or laboratory test abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results, and in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
17. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or patients who are Pfizer employees, including their family members, directly involved in the conduct of the study.
18. Fertile male patients or female patients of childbearing potential who are unwilling or unable to follow contraceptive requirements.
19. Pregnant or breastfeeding women.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Phase 2 open-label, randomized: Event-free survival (EFS) based on Investigator assessment. | Baseline to Month 24.
  EFS is defined as the time from randomization until first event (ie, progression, recurrence following response, second malignancy or death without progression or recurrence).
Phase 1: First Cycle Dose-Limiting Toxicities (DLT) | First cycle (cycle length is approximately 21 days)
  For Dose Escalation/Determination Part: DLT defined as any of the following events occurring during the first treatment cycle and considered at least possibly-related to study medication:Grade 4 neutropenia lasting greater than 7 days;Grade 4 thrombocytopenia lasting greater than 7 days or need for platelet transfusion for a platelet count of < 20,000 per cubic millimeters twice within a 7-day period;greater than 14-day delay in the start of a subsequent course because of neutropenia or thrombocytopenia;Grade 3 or greater non-hematologic toxicities despite optimal treatment;any Grade 2 or greater non-hematologic toxicity requiring discontinuation or interruption of palbociclib for 7 or more consecutive days during the first cycle or any grade non-hematologic toxicity that delays the start of Cycle 2 by more than 14 days;clinically significant non-hematologic laboratory test abnormality Grade 3 or greater not resolving to Grade 1 or baseline within 7 days.
Phase 1: Dose Expansion Parts: Frequency of adverse events | At least 28 days after last dose
  For Dose Expansion and Tumor-Specific Expansion Parts: Adverse events to be reported during treatment and for at least 28 days after last dose.
Phase 1: Dose Expansion Parts: Percentage of Participants With Complete Response or Partial Response | Through the end of treatment (up to at least 28 days after last dose)
  For Dose Expansion and Tumor-Specific Expansion Parts: patients with confirmed Complete Response or Partial Response per Response Evaluation Criteria in Solid Tumors (RECIST, v.1.1) or modified Response Assessment in Neuro-Oncology (RANO) for central nervous system malignancies, or International Neuroblastoma Response Criteria (INRC) for neuroblastoma, during study treatment, assessed approximately every 2 to 4 cycles (each cycle is approximately 21 days).

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Frequency of adverse events | At least 28 days after last dose
  Adverse events to be reported during treatment and for at least 28 days after last dose.
Phase 1 and Phase 2: Percentage of participants with laboratory abnormalities | At least 28 days after last dose
  Magnesium, Calcium, Creatinine, Albumin, Alanine aminotransferase, Aspartate aminotransferase, Glucose, Phosphorus, Total Bilirubin, Blood urea nitrogen, Alkaline phosphatase, Sodium, Potassium, Chloride, Platelet Count, White Blood Cell Count (differential), hemoglobin, INR or prothrombin Time, HbA1c
Phase 1 and Phase 2: Number of Participants With Clinically Significant Treatment-emergent Electrocardiogram (ECG) Findings | At least 28 days after last dose
  Clinically significant ECG findings included: corrected QT (QTc) > 450 ms, QTc >500 ms, change in QTc between 30 and 60 ms, change in QTc greater than or equal to 60 ms.
Phase 1 and Phase 2: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | At least 28 days after last dose
  systolic and diastolic blood pressure, pulse
Phase 2 open-label, randomized: Event-free survival (EFS) assessed by an independent review committee. | Baseline to Month 24.
  EFS is defined as the time from randomization until first event (ie, progression, recurrence following response, second malignancy or death without progression or recurrence).
Phase 1 and Phase 2: Percentage of Participants With Complete Response or Partial Response | Through the end of treatment (up to at least 28 days after last dose)
  Patients with confirmed Complete Response or Partial Response per Response Evaluation Criteria in Solid Tumors (RECIST, v.1.1) or modified Response Assessment in Neuro-Oncology (RANO) for central nervous system malignancies, or International Neuroblastoma Response Criteria (INRC) for neuroblastoma, during study treatment, assessed approximately every 2 to 4 cycles (each cycle is approximately 21 days).
Phase 1 and Phase 2: Duration of response (DoR) for Participants Who Achieved Complete Response or Partial Response | Up to 2 years
  DoR defined as time from date of first response (Complete Response or Partial Response) in responders to date of progression or death
Phase 1 and Phase 2: Progression Free Survival (PFS) | Up to 2 years
  PFS defined as time from date of enrollment to earliest date of the death or progressive disease
Phase 1 and Phase 2: Overall Survival (OS) | Up to 2 years
  OS defined as the time from enrollment to date of death due to any cause.
Phase 2 : comparison of PET-CT response assessment to objective response on CT/MRI. | up to completion of Cycle 4 ( 12 weeks of therapy)
  PET-CT response assessment will be compared to objective response on MRI/CT, as data permit.
Phase 2: the impact of the combination of palbociclib with TMZ and IRN treatment on the quality of life (QoL) of patients with refractory or recurrent EWS. | Up to Cycle 5 (completion of 12 weeks of treatment)
  Results of QoL reported by patient at baseline and after 2 and 4 cycles using age-appropriate PROMIS tools will be summarized for both treatment arms, as data permit.
  Days of hospitalization will be compared in both treatment arms.
Phase 1 and Phase 2:Palbociclib Pharmacokinetics, Maximum observed plasma concentration during a dosing interval at steady state (Css, max) | PK sampling at time points during Cycle 1 (day 2, 5, 6, 14) and Cycle 2 (day 5 and 14). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Palbociclib Pharmacokinetics, Maximum plasma concentration time (Tmax) | PK sampling at time points during Cycle 1 (day 2, 5, 6, 14) and Cycle 2 (day 5 and 14). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Palbociclib Pharmacokinetics, Area under the concentration-time curve during a dosing interval at steady state (AUCss,t) | PK sampling at time points during Cycle 1 (day 2,5, 6,14) and Cycle 2 (day 5 and 14). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Palbociclib Pharmacokinetics, Measured concentration at the end of a dosing interval at steady state (taken directly before next administration) (Css,trough) | PK sampling at time points during Cycle 1 (day 2, 5, 6, 14) and Cycle 2 (day 5 and 14). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Palbociclib Pharmacokinetics, Oral plasma clearance (CL/F) | PK sampling at time points during Cycle 1 (day 2, 5, 6, 14) and Cycle 2 (day 5 and 14). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Temozolomide Pharmacokinetics, Maximum observed plasma concentration during a dosing interval at steady state (Css, max) | PK sampling at time points during Cycle 1 (day 5) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Temozolomide Pharmacokinetics, Maximum plasma concentration time (Tmax) | PK sampling at time points during Cycle 1 (day 5) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Temozolomide Pharmacokinetics, Area under the concentration-time curve during a dosing interval at steady state (AUCss,t) | PK sampling at time points during Cycle 1 (day 5) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Temozolomide Pharmacokinetics, Measured concentration at the end of a dosing interval at steady state (taken directly before next administration) (Css,trough) | PK sampling at time points during Cycle 1 (day 5) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Temozolomide Pharmacokinetics, Oral plasma clearance (CL/F) | PK sampling at time points during Cycle 1 (day 5) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Irinotecan (and active metabolites) Pharmacokinetics, Maximum observed plasma concentration during a dosing interval at steady state (Css, max) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Irinotecan (and active metabolites) Pharmacokinetics, Maximum plasma concentration time (Tmax) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Irinotecan (and active metabolites) Pharmacokinetics, Area under the concentration-time curve during a dosing interval at steady state (AUCss,t) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Irinotecan (and active metabolites), Measured concentration at the end of a dosing interval at steady state (taken directly before next administration) (Css,trough) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1 and Phase 2: Irinotecan (and active metabolites) Pharmacokinetics, Oral plasma clearance (CL/F) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Topotecan (and active metabolites) Pharmacokinetics, Oral plasma clearance (CL/F) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Topotecan (and active metabolites), Measured concentration at the end of a dosing interval at steady state (taken directly before next administration) (Css,trough) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Topotecan (and active metabolites) Pharmacokinetics, Area under the concentration-time curve during a dosing interval at steady state (AUCss,t) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Topotecan (and active metabolites) Pharmacokinetics, Maximum plasma concentration time (Tmax) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Topotecan (and active metabolites) Pharmacokinetics, Maximum observed plasma concentration during a dosing interval at steady state (Css, max) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Cyclophosphamide Pharmacokinetics, Oral plasma clearance (CL/F) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Cyclophosphamide Pharmacokinetics, Maximum observed plasma concentration during a dosing interval at steady state (Css, max) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Cyclophosphamide Pharmacokinetics, Maximum plasma concentration time (Tmax) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Cyclophosphamide Pharmacokinetics, Area under the concentration-time curve during a dosing interval at steady state (AUCss,t) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit
Phase 1: Cyclophosphamide Pharmacokinetics, Measured concentration at the end of a dosing interval at steady state (taken directly before next administration) (Css,trough) | PK sampling at time points during Cycle 1 (day 2, 5 and 6) and Cycle 2 (day 5). Each cycle is 21 days.
  Multiple Dose (assuming steady state is achieved), as data permit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (99):
- United States (63):
  - University of Alabama at Birmingham/Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - MemorialCare Health System - Long Beach Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - UCSF Medical Center, San Francisco, California
  - University of California San Francisco,, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins All Children's Outpatient Care Center, St. Petersburg, Florida
  - Johns Hopkins All Children's Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Medical Office Building, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Novak Center for Children's Health, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - John R. Oishei Childrens Hospital, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Morgan Stanley Children's Hospital of New York-Presbyetrian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Cincinnati Children's Liberty Campus, Liberty Township, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Children's Hospital and Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Buerger Center for Advanced Pediatric Care, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Blood and Cancer Center, Austin, Texas
  - Dell Children's Medical Center, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Cook Children's H/O Infusion Center, Grapevine, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Medical Center Plano, Plano, Texas
  - Intermountain - Primary Children's Hospital, Salt Lake City, Utah
  - Primary Children's Hospital Outpatient Services, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Brazil (6):
  - Hospital Pequeno Principe / A ssociacao Hospitalar de Protecao a Infancia, Curitiba, Paraná
  - Hospital Pequeno Príncipe, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Hospital Santa Marcelina, São Paulo
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Czechia (2):
  - Detska nemocnice FN Brno, Brno, Brno-město
  - Fakultni nemocnice v Motole, Prague, Praha 5
- France (4):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Gustave Roussy, Villejuif, Val-de-marne
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille
- Universitätsklinikum Essen, Essen, North Rhine-Westphalia, Germany
- India (3):
  - Artemis hospital, Gurugram, Haryana
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
- Instytut Matki i Dziecka, Warsaw, Masovian Voivodeship, Poland
- Slovakia (2):
  - Detska fakultna nemocnica s poliklinikou Banska Bystrica, Banská Bystrica
  - Narodny ustav detskych chorob, Bratislava
- South Korea (4):
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Comunidad de
- Sahlgrenska Universitetssjukhuset Östra, Gothenburg, Västra Götalands LÄN [se-14], Sweden
- Turkey (Türkiye) (2):
  - Ege Universitesi Hastanesi, Izmir, İ̇zmir
  - Hacettepe Universite Hastaneleri, Ankara
- United Kingdom (4):
  - Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Royal Hospital for Children, Glasgow, Scotland
  - Leeds General Infirmary, Leeds
  - University College London Hospital, NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481092